CLINICAL TRIAL: NCT00419016
Title: Association Between Schizophrenia and Cancer
Status: Completed | Type: Observational
Sponsor: Sheba Medical Center (Other Government)
Other Study IDs: SHEBA-06-4489-RG-CTIL
Record Dates: First submitted 2007-01-04; First posted 2007-01-05 (Estimated); Last update posted 2007-01-05 (Estimated); Status verified 2007-01

CONDITIONS: Schizophrenia; Cancer
MeSH Terms: conditions — Schizophrenia; Neoplasms

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
A family study of the negative association betweeen schizophrenia and cancer

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gilad Gal, PhD, Principal Investigator — The Gertner Institute